CLINICAL TRIAL: NCT04569149
Title: Primordial Dwarfism Registry at Nemours Children's Hospital, Delaware
Brief Title: Primordial Dwarfism Registry
Status: Recruiting | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Potentials Foundation (Unknown); Walking with Giants Foundation (Unknown)
Responsible Party: Principal Investigator, Angela Duker, Genetic Counselor/Coordinator of Skeletal Dysplasia Program, Nemours Children's Clinic
Other Study IDs: MB001
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: MOPDII; Meier-Gorlin Syndrome; Saul-Wilson Syndrome; Microcephalic Primordial Dwarfism; IMAGe Syndrome; RNU4atac-opathy (e.g MOPDI, Lowry-Wood Syndrome, and Roifman Syndrome); LIG4 Syndrome
Keywords: microcephalic primordial dwarfism
MeSH Terms: conditions — Microcephalic Osteodysplastic Primordial Dwarfism, Type II; Meier-Gorlin syndrome; Seckel syndrome 1; Intrauterine Growth Retardation, Metaphyseal Dysplasia, Adrenal Hypoplasia Congenita, And Genital Anomalies; Lowry Wood syndrome; Roifman syndrome; LIG4 Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this registry is to collect information on individuals with forms of microcephalic primordial dwarfism as well as related conditions. The study team hopes to learn more about these conditions and improve the care of people with them by establishing this registry.

DETAILED DESCRIPTION:
The registry will enable detailed natural history studies of various forms of microcephalic primordial dwarfism as well as related conditions. The study team hopes that identification of risk factors will allow for preventative treatments and thus a better quality of life for individuals with these diagnoses.

This study is limited to chart review, after signed informed consent obtained. There will be no additional visits or time in clinic because of participation in this registry. This study involves only the collection and storage of data extracted from the medical record. Records that may be requested and reviewed as a part of this study include but may not be limited to: specialist evaluations, surgical reports, results of blood and urine tests, genetic testing, x-rays, CT/MRI/MRA imaging. There are no special procedures, visits, or expectations of the individual as a result of participation in this registry. No one will be asked to have any specific testing for the sole purposes of this research.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with MOPDII, Meier-Gorlin syndrome, IMAGe syndrome, RNU4atac-opathies (MOPDI/III, Roifman syndrome, Lowry-Wood syndrome), LIG4 syndrome, and other classified as well as unclassified types of microcephalic primordial dwarfism and related conditions, as diagnosed by a medical provider, are eligible for this registry.

Exclusion Criteria:

* individuals without microcephalic primordial dwarfism or closely related conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any individual at any age with microcephalic primordial dwarfism or a closely related condition
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-03-11 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of the natural history of various forms of primordial dwarfism | 5 years
  Data will be collected at enrollment, and over time, to allow for analysis of associated concerns throughout the lifespan

CONTACTS AND LOCATIONS:
Overall Officials: Angela Duker, MS, Principal Investigator — Nemours
Locations (1):
- Nemours, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No